CLINICAL TRIAL: NCT00322751
Title: Phase I Study of Concurrent Radiotherapy With Weekly Topotecan for Primary Treatment of Inoperable Localized Non-small Cell Lung Cancer (NSCLC) (Stage I to IIIA)
Brief Title: Concurrent Radiotherapy With Weekly Topotecan for Primary Treatment of Inoperable Localized Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Dennie Jones, MD; Principal Investigator, University of New Mexico - CRTC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0529C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2009-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan — The starting dose for the first cohort will be 2 mg/m2/week. Increment between cohorts will be by 1 mg/m2/week if no toxicity related to topotecan occurs. All members of a dose cohort must have safely completed all radiotherapy and topotecan dosing prior to beginning enrollment in the next higher dose cohort. Increments will be reduced to 0.5 mg/m2 if mild to moderate toxicity occurs (grades 1 or 2). The escalation will continue until the maximum dose of 4 mg/m2/week is reached. Therefore the minimum number of dose levels (cohorts) is 3 to reach the goal of 4 mg/m2/week, and the maximum is 5.

SUMMARY:
Given the activity of single-agent Topotecan in NSCLC, there is both scientific rationale and a medical interest in studying this agent in combination with radiation. In addition, Topotecan administered on a weekly basis offers advantages over the daily x 5 regimen, i.e., the convenience of administration and fewer visits to the clinic.

DETAILED DESCRIPTION:
This is a study of chemoradiation for patient with inoperable non small cell lung cancer with poor pulmonary function. These patients have usually very limited treatment options because of the compromised lung function. Chemoradiation is usually superior to radiation alone, but has not been extensively tested in this patient population. Topotecan is a drug approved for lung cancer that has synergistic activity with radiation. The study will determine what is the safest dose of topotecan to use with radiation in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven non-small cell lung cancer Stage I to IIIA.
* Inoperable lung cancer because of poor respiratory lung function, or other medical reasons, as determined by the thoracic surgeon.
* PS < 2
* Age > 18 years
* Life expectancy of > 12 weeks
* Normal hematologic, liver, and renal function
* No metastatic disease as determined by CT-PET scanning and bone scan.
* No brain metastasis by MRI
* No contraindication to radiotherapy

Exclusion Criteria:

* Patients with uncontrolled CNS metastases.
* Active systemic infection.
* Serious, uncontrolled intercurrent medical or psychiatric illness.
* Secondary active primary malignancy.
* Inability to comply with requirements of the study.
* Any metastases outside of the mediastinum
* Histologically positive pleural or pericardial effusion
* Any chemotherapy within five years prior to enrollment on this protocol
* Prior radiotherapy administered to the chest
* Women who are pregnant or lactating
* FEV1 < 1 liter/minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the establishment of the maximum tolerated dose (MTD) of topotecan given weekly with RT | Treatment with topotecan will last until RT is completed. Treatment will stop if there is disease progression or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Dennie Jones, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States